CLINICAL TRIAL: NCT05636319
Title: A Randomized, Double-blind, Placebo-controlled Clinical Study to Evaluate the Efficacy, Safety, and Immunogenicity of SARS-CoV-2 Variant (BA.4/5) mRNA Vaccine (ABO1020) in Healthy Subjects Aged 18 Years and Older Who Have Completed the Full Vaccination
Brief Title: A Study to Evaluate the Efficacy, Safety, and Immunogenicity of SARS-CoV-2 Variant (BA.4 /5) mRNA Vaccine
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Suzhou Abogen Biosciences Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: ABO1020-301
Record Dates: First submitted 2022-11-23; First posted 2022-12-05 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2023-09

CONDITIONS: COVID-19
Keywords: COVID-19; Omicron
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Phase1/2: 30 subjects will be randomized in a ratio of 2:1 to receive ABO1020 and placebo, intramuscularly injected in the lateral deltoid region of the upper arm according to the two doses immunization schedule on Day 0 and Day 28.
  Phase3: 15000 subjects will be randomized in a ratio of 1:1 to receive ABO1020 and placebo, intramuscularly injected in the lateral deltoid region of the upper arm according to the two doses immunization schedule on Day 0 and Day 28.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group 1: ABO1020 (Experimental): Intramuscularly inject 15 μg of ABO1020 into lateral deltoid region of the upper arm of subjects on D0 and D28, respectively.
  Interventions: Biological: ABO1020
- Test group 2: Placebo (Placebo Comparator): Intramuscularly inject 0 μg of placebo into lateral deltoid region of the upper arm of subjects on D0 and D28, respectively.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: ABO1020 — Vaccine
  Arms: Test group 1: ABO1020
Biological: Placebo — Placebo
  Arms: Test group 2: Placebo

SUMMARY:
A Randomized, Double-blind, Placebo-controlled Clinical Study to Evaluate the Efficacy, Safety, and Immunogenicity of SARS-CoV-2 Variant (BA.4 /5) mRNA Vaccine (ABO1020) in Healthy Subjects Aged 18 Years and Older Who Have Completed the Full Vaccination

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign the ICF approved by the Ethics Committee before any study procedure and agree to participate in the study.
2. Healthy male or female able to provide legal identity certificate and aged 18 years and older when signing the ICF.
3. Subjects who have previously been fully vaccinated either by 2 or 3 doses of SARS-CoV-2 inactivated vaccine. The last dose of immunization should be >6 months before administration of the investigational products.
4. Be able to communicate well with the investigator, and to understand and comply with the requirements of this clinical trial.
5. Males and females with childbearing potential voluntarily take effective contraceptive methods from signing ICF to 3 months after completing the vaccination, including sexual abstinence or effective contraceptive measures (e.g., intrauterine or implanted contraceptive device, oral contraceptives, injected or implanted contraceptives, sustained-release topical contraceptives, intrauterine device [IUD], condoms [male], diaphragm, and cervical cap).

Exclusion Criteria:

1. Positive SARS-CoV-2 rapid test at screening.
2. Prior medical history of severe acute respiratory syndrome (SARS), middle east respiratory syndrome (MERS).
3. Fever (axillary temperature or equivalent ≥ 37.3℃*) on the day of vaccination with this investigational vaccine or within recent 72 hours.
4. Abnormal vital signs (pulse < 60 bpm or > 100 bpm, systolic blood pressure ≥ 140 mmHg or diastolic blood pressure ≥ 90 mmHg when keeping awake) with clinical relevance.
5. Do not remain overall healthy (i.e., has medically deteriorated significantly since receiving the two-dose vaccination, is anticipated to have fatal outcome of uncontrolled diseases within 12 months, and is not able to provide blood as specified by the trial with anticipated, deleterious medical consequences) in the clinical judgment of the investigator based on medical history and physical examination.
6. Pregnant or lactating women, or those who plan to donate sperm or egg during the trial.
7. Prior history of allergic reaction or anaphylaxis to any vaccine or its excipients, e.g., hypersensitivity, urticaria, serious eczema, dyspnea, laryngeal edema, and angioedema etc.
8. Prior use of any other vaccine within 28 days before using the investigational products or planning to use any vaccine other than the investigational products during the study period.
9. Participation in the studies of any other interventional device or drug within 30 days before the screening, or current treatment with other investigational drug(s) or within 5 half-lives after taking the last dose of the study drug.
10. Hereditary hemorrhagic tendency or coagulation dysfunction (e.g., cytokine defects, coagulation disorders or platelet disorder), or a history of serious bleeding, or a history of massive bleeding after intramuscular injection or intravenous puncture or ecchymosis.
11. Known medical history or diagnosis confirming that subjects have diseases affecting immune system function, including cancer (except skin basal cell carcinoma), congenital or acquired immunodeficiency (e.g., infection with human immunodeficiency virus [HIV]), and uncontrolled autoimmune disease.
12. Serious or uncontrolled respiratory system disorders, cardiovascular disorders, nervous system disorders, blood and lymphatic system disorders, liver and kidney disorders, metabolism and skeletal disorders,etc. influencing study results evaluation at the investigator's discretion.
13. Asplenia or functional asplenia.
14. Long-term use (continuous use ≥14 days) of immunosuppressants or other immunomodulators (e.g., glucocorticoids: prednisone or similar drugs) within 6 months prior to administration of this investigational vaccine, except for topical medications (e.g., ointments, eye drops, inhalants or nasal sprays). And the topical medications should not exceed the recommended dose in the labels for use or induce any signs of systemic exposure.
15. Having received immunoglobulins and/or blood products within 3 months prior to administration of this investigational vaccine.
16. Suspected or known alcohol dependency or drug abuse, which may affect safety evaluation or subject's compliance at the investigator's discretion.
17. Planning to permanently move from the local area before study completion or leave the local area for a long time during the period of study visits.
18. Receiving antituberculosis treatment.
19. Staff of study site, sponsor and contract research organization (CRO) taking part in the study.
20. Other conditions that the investigators consider unsuitable for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14168 (Actual)
Dates: Start 2022-11-23 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
In Phase 1/2, Incidence of solicited adverse events | 0 to 14 days after each dose
  Solicited adverse events 0 to 14 days after each dose
In Phase 1/2, Incidence of unsolicited adverse events | 0 to 28 days after each dose
  Unsolicited adverse events 0 to 28 days after each dose
In Phase 3, efficacy after the second dose | 14 days after second dose
  Confirmed COVID-19 cases occurring from 14 days after the second dose

SECONDARY OUTCOMES:
In Phase 1/2, titer of Anti-SARS-CoV-2 live virus neutralizing antibody | 28 days after each dose and the corresponding ratio against Day 0 before the vaccination.
  Evaluate the immunogenicity of ABO1020
In Phase 1/2, Observation of Long-term Safety | 12 months after each dose
  Serious adverse events, adverse events of special interest and other medically attended adverse events through 12 months after each dose.
In Phase 3, titer of Anti-SARS-CoV-2 live virus neutralizing antibody | 28 days after each dose, 90 days and 180 days after the second dose and the corresponding ratio against Day 0 before the vaccination.
  Evaluate the immunogenicity of ABO1020
In Phase 3, Observation of long-term Safety | 12 months after each dose
  Serious adverse events, adverse events of special interest through 12 months after each dose.

CONTACTS AND LOCATIONS:
Locations (25):
- Indonesia (5):
  - RS Universitas Indonesia, Depok
  - RS YARSI, Jakarta
  - RSIJ Cempaka Putih, Jakarta
  - RSUP Persahabatan, Jakarta
  - Rumah Sakit Umum Pusat Nasional Dr. Cipto Mangunkusumo, Jakarta
- Pakistan (8):
  - Central Hospital, Gujranwala, Gujranwala
  - Maroof International Hospital, Islamabad, Islamabad
  - Rehman Medical Institute, Khaibar
  - Akram Medical Complex, Lahore
  - Avicenna Medical College, Lahore
  - Central Park Teaching Hospital, Lahore
  - National Hospital and Medical center, Lahore
  - Al-Shifa Trust Eye Hospital, Rawalpindi
- Philippines (8):
  - Manuel J. Santos Hospita, Butuan
  - Premiere Medical Center, Cabanatuan City
  - Silang Medical Center, Cavite
  - Davao Medical School Foundation, Davao City
  - St. Paul's Hospital Iloilo, Iloilo City
  - Healthcube Medical Clinic, Mandaluyong
  - Medical Center Manila, Manila
  - Philippine General Hospital, Manila
- United Arab Emirates (4):
  - Burjeel Medical City, Abu Dhabi
  - Life Care Hospital, Abu Dhabi
  - Medeor hospital, Abu Dhabi
  - AI Kuwait Hospital, Dubai

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hannawi S, Wu XH, Villalobos RE, Burhan E, Lallaine Borra MD, Gupta RK, Aquitania GP, Ang BWC, Mae A Zabat G, Roa CC Jr, Zoleta-De Jesus L, Yu DD, Wang M, Wu Y, Song WJ, Ying B, Qin CF. Efficacy, immunogenicity, and safety of a monovalent mRNA vaccine, ABO1020, in adults: A randomized, double-blind, placebo-controlled, phase 3 trial. Med. 2024 Oct 11;5(10):1282-1292.e3. doi: 10.1016/j.medj.2024.06.013. Epub 2024 Jul 17. PMID 39025066
- See also: Efficacy, immunogenicity, and safety of a monovalent mRNA vaccine, ABO1020, in adults: A randomized, double-blind, placebo-controlled, phase 3 trial, Med (2024), https://doi.org/10.1016/j.medj.2024.06.013 — https://doi.org/10.1016/j.medj.2024.06.013
- See also: Efficacy, immunogenicity, and safety of a monovalent mRNA vaccine, ABO1020, in adults: A randomized, double-blind, placebo-controlled, phase 3 trial, Med (2024), https://doi.org/10.1016/j.medj.2024.06.013 — https://pubmed.ncbi.nlm.nih.gov/39025066/